CLINICAL TRIAL: NCT03054454
Title: A Podiatry-led Multidisciplinary Intervention to Reduce the Burden of Foot Disease in People With Diabetes and End-stage Kidney Failure
Brief Title: A Podiatry Led MDT Intervention to Reduce the Burden of Foot Disease in Patients With End Stage Kidney Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South Tees Hospitals NHS Foundation Trust (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20720171
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus; Endstage Renal Disease
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Active Comparator): This group will receive Podiatry treatment and care from the MDT which is the intervention group.
  Interventions: Procedure: Podiatry
- comparator (No Intervention): This group will receive usual care

INTERVENTIONS:
Procedure: Podiatry — Podiatry treatments and care from the multidisciplinary team.
  Arms: intervention

SUMMARY:
Observational studies clearly show that people with diabetes and end-stage kidney failure have an increased risk of foot ulceration and leg amputation. However, there is very little evidence on addressing this problem.

Diabetes foot care teams have been shown to reduce hospital admissions, length of stay and leg amputation in people with diabetes. Since their introduction at The James Cook University Hospital (JCUH) major diabetes-related leg amputation rates have fallen by 86 percent (1995 to 2010).

People with diabetes and end-stage kidney failure require haemodialysis (blood cleaning) 3 times per week for several hours each time. This time commitment makes it difficult to attend other clinical appointments. An audit at JCUH shows that this population fails to attend the normal diabetes foot services.

This project aims to reduce the incidence of foot disease in people with diabetes and end-stage kidney failure on dialysis. The investigators will set up a podiatry-led intervention within the dialysis unit to prevent and promptly treat foot disease in this population. This will involve foot risk assessment, risk reduction and treatment during dialysis. The intervention will involve diabetes consultants, podiatrists, vascular and orthopaedic surgeons . In this way the investigators hope to reduce leg amputation, hospital admission, procedures to unblock arteries and death in this high risk group.

The study will run in the dialysis unit at JCUH. Patients will be divided into two groups: those attending for dialysis on a Monday, Wednesday and Friday will form the treatment group and those attending on a Tuesday, Thursday and Saturday will continue to be managed as at present. The investigators will collect data from patient health care records looking in particular at leg amputations, hospital admissions due to foot problems, foot surgery and operations to unblock arteries.

DETAILED DESCRIPTION:
Diabetes is the largest cause of leg amputation and kidney failure; 15-20% of people with diabetes will have a foot ulcer in their lifetime, with 5-10% having an ulcer at any one time. The history of a foot ulcer in a person with diabetes increases the risk of leg amputation 2-3 fold. A person with diabetes is 23 times more likely to have a leg amputation than a person without diabetes.

The risk of having a foot ulcer is increased by another four times and the risk of leg amputation by a further eight times in people with diabetes and kidney failure on dialysis compared to those with diabetes and normal kidney function. Kidney failure in people with diabetes increased by 56% between 2006 and 2010.

Sixty per cent of people who have diabetes and a leg amputation will be dead within 5 years. Those with end stage kidney failure and a foot ulcer have an even bleaker outcome: only 50% will be alive in 2 years. This reduces to 26% following leg amputation.

An audit in 2014 of the patients attending the dialysis unit at the hospital showed that half had diabetes. Of these, half had had a foot ulcer at some point. Half of these had an ulcer at the time of the audit. Less than one quarter of those with a foot ulcer had been reviewed by the Diabetes Foot Team. National guidance states that all people with diabetes and a foot ulcer should be seen by a diabetes foot team within one working day of the ulcer being detected.

The investigators looked for evidence to show how to reduce the risk of foot problems in people with diabetes and end-stage kidney failure on dialysis but were unable to find any evidence.

Regional kidney and diabetes specialist groups have confirmed that there is no such work to address this problem anywhere in the North East and neither were aware of such an intervention anywhere in the UK.

None of the leading Consultants in the UK working in the field of diabetes-foot disease are aware of the existence of a project like this but were in agreement about the need for one.

The existing literature shows the severity of the problem but not the solution. The investigators plan to provide evidence to show an effective and cost-saving solution to reduce the burden of diabetic foot disease in people with diabetes and end-stage kidney failure People who require dialysis attend the dialysis unit 3 times a week on fixed days and in a fixed session which doesn't tend to change. People with diabetes and kidney failure on dialysis will be divided into 2 groups: a treatment group and a comparator group. The treatment group will be those that have dialysis on a Monday, Wednesday and Friday. The comparator group will be those who have dialysis on a Tuesday, Thursday and Saturday

The comparator group will continue to receive diabetes foot care using the standard model that is in existence at present (i.e. screening at GP practice, podiatry review close to home and referral to a hospital diabetes foot team when necessary)

The treatment group will be reviewed by a podiatrist while they are having dialysis. The Podiatrist will examine their feet at the first meeting and look for diabetic foot problems, if not present, make a standard assessment of the risk of diabetic foot problems developing. Further management will be guided by this assessment.

The population will fall into two groups :those without active foot problems but at high risk of developing foot problems; and those with active foot disease (e.g. foot ulcer). High risk patients without current foot problems will receive a package of treatments aimed at preventing foot ulcers (including education, removal of hard skin, foot and nail care, changes to shoes and the provision of bespoke insoles, creams and further podiatric review.

Those with active foot problems will have investigations and treatment according to individual need, which might include x-rays, tests for bacterial infection, blood tests, removal of hard skin, wound dressings and offloading. Treatments to improve blood supply to the feet and surgical removal of infected tissue might be needed. This will be lead by the podiatrist. However, other members of the diabetes foot care team (MDT) will be involved as required, using the existing weekly diabetes foot MDT meetings as a forum for discussion of the patients. Other MDT members will then also see the patients on the dialysis unit, thus providing patient-centred care.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Type 1 2, secondary or MODY
* End-stage renal failure (CKD stage 5)
* Routinely attending the dialysis unit at The James Cook University Hospital for regular dialysis

Exclusion Criteria:

* Lack of capacity
* Bilateral lower limb amputees
* People on dialysis who do not have diabetes

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Nights spent in hospital with a diabetes-related foot problem. | 1 year
  Nights spent in hospital with a diabetes-related foot (below ankle) problem (ulceration, cellulitis, foot pain, swelling, foot infection/ osteomyelitis, necrosis, gangrene, blister, ischaemia, fracture)

SECONDARY OUTCOMES:
number of below knee amputations attributed to diabetic foot disease | 1 year
  the no. of below knee amputations will be recorded in this group and compared tot he comparator group who will receive usual care

CONTACTS AND LOCATIONS:
Overall Officials: Simon Ashwell, Dr, Principal Investigator — Trust consultant

IPD SHARING:
Plan to Share IPD: No